CLINICAL TRIAL: NCT02522325
Title: Behavioral Effects of Drugs (Inpatient): 31 (Cocaine and Phendimetrazine)
Brief Title: Reinforcing Effects of Cocaine During Phendimetrazine Maintenance
Acronym: BED IN 31
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 15-0553; R01DA036553 (NIH)
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — phendimetrazine; Cocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be maintained on oral placebo, administered twice daily for approximately two weeks. Cocaine will be administered acutely during placebo maintenance. Placebo will be administered acutely during placebo maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo
- Phendimetrazine (Experimental): Subjects will be maintained on oral phendimetrazine (up to 210 mg/day) administered twice daily for approximately two weeks. Cocaine will be administered acutely during placebo maintenance. Placebo will be administered acutely during placebo maintenance.
  Interventions: Drug: Phendimetrazine; Drug: Cocaine

INTERVENTIONS:
Drug: Phendimetrazine — Phendimetrazine will be administered in divided doses twice daily.
  Other Names: Bontril
  Arms: Phendimetrazine
Drug: Cocaine — Intranasal cocaine will be administered during experimental sessions.
Drug: Placebo — Placebo capsules will contain only cornstarch.
  Arms: Placebo

SUMMARY:
This study will determine the initial efficacy of phendimetrazine as a pharmacotherapy for cocaine dependence. A rigorous, inpatient human laboratory study will be conducted in which the subjective, physiological and reinforcing effects of cocaine are evaluated during maintenance on placebo and phendimetrazine.

ELIGIBILITY:
Inclusion Criteria:

* Recent cocaine use

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance abuse or dependence that are deemed by the study physicians to interfere with study completion
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation
* Females not currently using effective birth control
* Contraindications to cocaine or phendimetrazine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky Department of Behavioral Science, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty subjects were enrolled, but one was removed from the study due to an adverse event, leading to 29 completers.
Groups:
- Placebo First, Then Phendimetrazine: Subjects were maintained on placebo for approximately 2 weeks, then they were crossed over to 210 mg phendimetrazine daily for approximately 2 weeks.
- Phendimetrazine First, Then Placebo: Subjects were maintained on 210 mg phendimetrazine for approximately 2 weeks, then they were crossed over to placebo daily for approximately 2 weeks.
Period: Overall Study
Arm/Group | Placebo First, Then Phendimetrazine | Phendimetrazine First, Then Placebo
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Completers: Baseline demographics for study completers
Arm/Group | Study Completers
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Times Cocaine Was Selected in the Presence of a Monetary Reward Alternative
Description: The reinforcing effects of cocaine were determined using a modified progressive ratio procedure in which subjects made 10 choices between a portion of each available cocaine dose and money (US$0.25). Reinforcing effects are measured for each cocaine dose during both phendimetrazine and placebo maintenance.
Time Frame: After at least seven days of maintenance placebo or target phendimetrazine dose
Measure: Mean (Standard Error); unit: Cocaine Choices
Groups:
- Placebo: Subjects were maintained on Placebo for at least 7 days.
- Phendimetrazine: Subjects were maintained on 210 mg Phendimetrazine for at least 7 days.
Arm/Group | Placebo | Phendimetrazine
Number analyzed (Participants) | 29 | 29
Cocaine Choices
  0 mg Cocaine | .34 (.34) | .24 (.15)
  20 mg Cocaine | 4.31 (.81) | 3.9 (.85)
  40 mg Cocaine | 4.69 (.89) | 3.83 (.85)
  80 mg Cocaine | 5.90 (.8) | 5.03 (.87)

ADVERSE EVENTS:
Time Frame: Approximately 1 month of inpatient admission
Groups:
- Placebo: Subjects were maintained on placebo for approximately 2 weeks.
- Phendimetrazine: Subjects were maintained on 210 mg phendimetrazine for approximately 2 weeks.
Arm/Group | Placebo | Phendimetrazine
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT02522325/Prot_SAP_000.pdf